CLINICAL TRIAL: NCT01384760
Title: A Randomized Controlled Study to Examine the Effect of Lifestyle Modification Program in Obstructive Sleep Apnea Patients
Brief Title: Lifestyle Modification Program to Treat Obstructive Sleep Apnea Patients
Acronym: OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Associate Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Resp/Ng/2011
Record Dates: First submitted 2011-06-10; First posted 2011-06-29 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle modification program (Active Comparator): At the 1st session, the dietitian carried out a complete behavioral assessment, with emphasis on patient's current eating and lifestyle patterns, specific eating-related behaviors, knowledge of risks associated with current eating patterns, and concerns and feelings about specific lifestyle changes. In the subsequent follow up visit, the dietitian reviewed the 7-day food diaries to ensure nutritional adequacy and treatment compliance, and also offered recommendations for controlling caloric intake.
  Patients were encouraged to see an exercise instructor who designed an individualized suitable exercise regime with cardiovascular and resistance exercises for the patients to perform at home. Subjects were encouraged to perform 30-minute aerobic exercise 2-3 times a week.
  Interventions: Behavioral: Lifestyle modification
- Simple lifestyle advice (Placebo Comparator): Subjects in control group received simple lifestyle advice from a clinician at baseline and month 6. This was a brief discussion about the general health risk associated with OSA and importance of balanced diet. Subjects were encouraged to perform regular 30-minute exercise 2 to 3 times per week. This was to resemble routine clinical practice.
  Interventions: Behavioral: Simple lifestyle advice

INTERVENTIONS:
Behavioral: Lifestyle modification — During the first 4 months, subjects will come for a counseling session weekly and then monthly for the following months. During each counseling session (15 to 20 minutes), the registered dietitian will review the seven-day food diaries and offer recommendations for controlling caloric intake. A varied balanced diet with an emphasis on fruit and vegetables, and low-fat and low calorific products in appropriate portions were encouraged. The registered dietitian will also review the daily activity log sheet to check the exercise adherence and progression set by exercise instructor. Subjects will be encouraged to do 30 minutes aerobic exercise two to three times a week.
  Other Names: Intervention group
  Arms: Lifestyle modification program
Behavioral: Simple lifestyle advice — Subjects in control group will receive simple lifestyle advice from a clinician at baseline and month 6. This will be a brief discussion about the general health risk associated with OSA and importance of balanced diet. Subjects are encouraged to perform regular 30-minute exercise 2 to 3 times per week. This is to resemble routine clinical practice.
  Other Names: Control group
  Arms: Simple lifestyle advice

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common form of sleep-disordered breathing (SDB) characterized by repetitive episodes of cessation of breathing during sleep due to upper airway collapse. It causes sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor quality of life. In addition, OSAS is associated with non-fatal and fatal cardiovascular consequences including sudden death, in addition to an increased risk of road traffic accidents. Continuous positive airway pressure (CPAP) is considered as the first-line treatment for OSA. Oral appliance has been shown to reduce the severity of sleep disordered breathing and leads to symptomatic improvement especially in mild to moderate OSA. The compliance with CPAP is low particularly in mild or moderate OSA patients and it is not a curative treatment of OSA. It has to be used in every night on a regular basis. Weight reduction has always been advocated in patients with OSA who are overweight and may lead to improvement in the severity of OSA. The existing studies about weight loss are limited by small sample size, short duration (<6 months), focus on very low calorie diet program or surgically induced weight loss program only. However, none of them have applied lifestyle modification program (LMP) which emphasizes on long term lifestyle and behavior change. Therefore, the investigators plan to conduct a randomized controlled trial among Chinese OSA patients by comparing the efficacy of LMP against usual clinical lifestyle advice alone on the improvement of OSA symptoms.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common form of sleep-disordered breathing (SDB) characterized by repetitive episodes of cessation of breathing during sleep due to upper airway collapse. It causes sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor quality of life. In addition, OSAS is associated with non-fatal and fatal cardiovascular consequences including sudden death, in addition to an increased risk of road traffic accidents.

OSAS is equally common among the middle-aged male Caucasian and Hong Kong (HK) Chinese populations with prevalence rates of at least 4%. The prevalence and severity of OSAS tend to increase through adult life, peaking in the late fifties to mid sixties, after which it fails to increase or decrease. Another group of investigators reported high prevalence rates of SDB in a group aged 65-95 years of 70% for men and 56% for women, at least double those reported for middle-aged cohorts.

Risk factors for OSA include obesity, increasing age, being male, abnormal craniofacial morphology, nasal obstruction, genetic factors. OSA is associated with several cardiovascular consequences and social consequences e.g. motor vehicle accidents, impaired cognitive performance, depression. Various epidemiologic studies have shown an association between OSA and hypertension. In cross-sectional study, OSA was associated with increased prevalence of self-reported heart failure and stroke. OSA has been shown to be independently associated with coronary artery disease after adjustment for traditionally considered risk factors.

Continuous positive airway pressure (CPAP) is considered as the first-line treatment for OSA. Oral appliance has been shown to reduce the severity of sleep disordered breathing and leads to symptomatic improvement especially in mild to moderate OSA. The compliance with CPAP is low particularly in mild or moderate OSA patients and it is not a curative treatment of OSA. It has to be used in every night on a regular basis. Weight reduction has always been advocated in patients with OSA who are overweight and may lead to improvement in the severity of OSA. A population-based longitudinal study showed that a 10% weight loss predicted a 26% decrease in apnoea-hypopnoea index (AHI), a count of the number of upper airway obstructions per hour of sleep.

The existing studies about weight loss are limited by small sample size, short duration (<6 months), focus on very low calorie diet program or surgically induced weight loss program only. However, none of them have applied lifestyle modification program (LMP) which emphasizes on long term lifestyle and behavior change. Therefore, the investigators plan to conduct a randomized controlled trial among Chinese OSA patients by comparing the efficacy of LMP against usual clinical lifestyle advice alone on the improvement of OSA symptoms.

Aim of the study:

The investigators aim to test the hypothesis that LMP is superior to lifestyle advice alone in the management of Chinese patients with OSA. The primary outcome measure is the change of AHI. The secondary outcome measures are changes in quality of life, symptoms related to OSA, glucose, and insulin metabolism parameters.

Hypothesis:

The investigators hypothesize that more OSA patients in a low glycemic index dietary intervention program than patients receiving simple lifestyle advice alone will have reduction in AHI.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 80 years
* AHI ≥ 5/hour
* Body mass index (BMI) greater than or equal to 25
* Written informed consent obtained

Exclusion criteria:

* Presence of sleepiness which may constitute risk to self or others
* Chronic kidney, thyroid, or liver disease
* Coexistence of sleep disorders other than OSA
* History of previous surgery to upper airway (except those for nasal problems)
* Previous surgical or current medical treatment for OSA Pregnant women

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna SS Ng, MBChB, Principal Investigator — Chinese Univesrity of Hong Kong; David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Ng SSS, Chan RSM, Woo J, Chan TO, Cheung BHK, Sea MMM, To KW, Chan KKP, Ngai J, Yip WH, Ko FWS, Hui DSC. A Randomized Controlled Study to Examine the Effect of a Lifestyle Modification Program in OSA. Chest. 2015 Nov;148(5):1193-1203. doi: 10.1378/chest.14-3016. PMID 25763792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 185 patients were screened and 104 underwent randomization
Period: Overall Study
Arm/Group | Lifestyle Modification Program | Simple Lifestyle Advice
Started | 61 | 43
Randomized | 61 | 43
Completed | 45 | 37
Not Completed | 16 | 6
Not completed — Lost to Follow-up | 0 | 6
Not completed — Protocol Violation | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Modification Program | Simple Lifestyle Advice | Total
Number analyzed (Participants) | 61 | 43 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.1) | 52 (9.3) | 51.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 48 | 30 | 78
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (3.9) | 30.5 (4.2) | 30.3 (4.0)
Neck circumference (cm) [Mean (Standard Deviation); unit: cm] | 39.9 (3.3) | 40.3 (3.7) | 40.1 (3.5)
smoking status [Number; unit: participants]
  never smoke | 44 | 31 | 75
  quitted smoking | 6 | 6 | 12
  current smoking | 11 | 6 | 17
AHI - events/hour [Mean (Standard Deviation); unit: events per hour] | 43.4 (20) | 42.5 (20) | 43 (19.8)
minSaO2 [Mean (Standard Deviation); unit: percentage] | 69.6 (9.7) | 65.1 (17.9) | 67.2 (10.2)
Score on Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) is a self-reporting questionnaire to assess subjective sleepiness and relies on dosing behavior in eight different situations of relatively low soporific nature, asking the respondent to rate the likelihood of falling asleep on a scale from 0 to 3, were 0 indicates no chance and 3 being the greatest chance of dosing. The scores for the eight questions are added together to obtain a single number.
  A number in the 0-9 range is considered to be normal while a number of >10 indicates pathological sleepiness.
  units on a scale | 11.4 (5.7) | 10.2 (4.7) | 11.0 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI) at One Year
Description: AHI is a count of the number of upper airway obstruction per hour of sleep. The index will be derived from the overnight home sleep study.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Lifestyle Modification Program | Simple Lifestyle Advice
Number analyzed (Participants) | 61 | 43
events per hour | 35.3 (21.7) | 39.6 (19.5)

2. Secondary Outcome: Epworth Sleepiness Score (ESS)
Description: The Epworth Sleepiness Scale (ESS) is a questionnaire for assessing daytime sleepiness. It was first described in 1991 as a simple, self-administered questionnaire. The questionnaire is based on eight common situations in life. Subjects are asked to rate on a scale of 0-3 about how likely they would fall asleep or doze off in these circumstances. This gives a total score of 0 to 24 in each subject.The total score ranges from 0 to 24, with higher scores indicating higher sleepiness.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Modification Program | Simple Lifestyle Advice
Number analyzed (Participants) | 61 | 43
units on a scale | 8.9 (4.8) | 9.2 (4.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Lifestyle Modification Program | Simple Lifestyle Advice
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No